CLINICAL TRIAL: NCT04167137
Title: A Phase 1, Open-label, Multicenter Study of SYNB1891 Administered by Intratumoral Injection to Patients With Advanced/Metastatic Solid Tumors and Lymphoma Alone and in Combination With Atezolizumab
Brief Title: Safety and Tolerability of SYNB1891 Injection Alone or in Combination With Atezolizumab in Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Synlogic (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYNB1891-CP-001
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Solid Neoplasm; Lymphoma
Keywords: solid tumor
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Dose-escalating, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: SYNB1891 Monotherapy (Experimental): SYNB1891 monotherapy was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles for up to 24 months/35 cycles. The starting dose of SYNB1891 in the first cohort was 1 × 10^6 live cells and was increased in approximately 3-fold increments in subsequent cohorts.
  Interventions: Drug: SYNB1891
- Arm 2: SYNB1891 in Combination with Atezolizumab (Experimental): SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles for up to 24 months/35 cycles. The dose of SYNB1891 in the first cohort was 1 × 10^7 live cells and was increased in an approximately 3-fold increment to 3 × 10^7 live cells in the second cohort.
  Atezolizumab was administered in accordance with its recommended dose and schedule (1200 mg IV Q3W) on Day 1 of each cycle for up to 24 months/35 cycles. On days when atezolizumab and SYNB1891 were both administered, SYNB1891 was administered first, followed by at least 1 hour of observation prior to the atezolizumab infusion.
  Interventions: Drug: SYNB1891; Drug: Atezolizumab

INTERVENTIONS:
Drug: SYNB1891 — SYNB1891 was administered as an IT injection over a dose range of 1 x 10^6 to 3 x 10^8 live cells in Arm 1 and 1 x 10^7 to 3 x 10^7 in Arm 2.
Drug: Atezolizumab — Atezolizumab was administered in accordance with its recommended dose and schedule (1200 mg IV Q3W).
  Arms: Arm 2: SYNB1891 in Combination with Atezolizumab

SUMMARY:
This Phase 1, open-label, multicenter, 2-arm study was designed to evaluate SYNB1891 when administered either as monotherapy (Arm 1) or in combination with atezolizumab (Arm 2) in participants with advanced/metastatic solid tumors or lymphoma. The primary objective was to evaluate the safety and tolerability of study treatment, with a secondary objective of assessing preliminary tumor response to treatment and exploratory objectives of evaluating the pharmacokinetics/pharmacodynamics (PK/PD) of study treatment.

DETAILED DESCRIPTION:
Arm 1 comprised intratumoral (IT) injections of SYNB1891 monotherapy to determine the single-agent maximum tolerated dose (MTD). The starting dose of SYNB1891 in the first cohort was 1 × 10^6 live cells and was increased in approximately 3-fold increments in subsequent cohorts until MTD determination in accordance with the modified toxicity probability interval (mTPI) algorithm (Ji et al 2013). Dose escalation was to proceed until the target dose-limiting toxicity (DLT) range (approximately 30%) for SYNB1891 monotherapy was determined based on DLTs observed in Cycle 1. The dose selected as achieving the target DLT range was to be considered the MTD. DLTs were defined in the protocol as certain treatment-related Grade 3/4 laboratory values, sepsis, toxicity resulting in death, discontinuation of Cycle 1, or delay of Cycle 2.

Arm 2 comprised IT injections of SYNB1891 combined with standard dose atezolizumab (1200 mg intravenously [IV] every 3 weeks [Q3W]). Arm 2 dosing began after all participants in Arm 1 Cohort 4 completed their Cycle 1 DLT safety evaluation. The starting dose of IT SYNB1891 in the first cohort of Arm 2 was at the SYNB1891 Arm 1 Cohort 3 dose level. SYNB1891 dosing in the Arm 2 cohorts increased in approximately 3-fold increments in subsequent cohorts until recommended Phase 2 dose (RP2D) determination. SYNB1891 combination dosing in Arm 2 was always at least 1 dose level below the SYNB1891 monotherapy dose being evaluated in Arm 1, with combination doses not escalated above the SYNB1891 single-agent MTD established in Arm 1.

In both arms, after an initial 4 cycles (21 days per cycle) of study treatment, participants who did not have progressive disease may have received additional cycles of their assigned study treatment for up to 24 months (i.e., Cycles 5 to 35) after the initial dose.

The maximum time of study participation for a participant may have been up to 26 months, including the screening period (up to 28 days), treatment administration period (up to 24 months), and Safety Follow-up period (30 ± 5 days after the last dose).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to voluntarily complete the informed consent process (participant or participant's representative).
2. Adults aged ≥ 18 years (on the day of signing informed consent) with histologically- or cytologically-confirmed stage III or IV advanced/metastatic solid tumor or lymphoma for which no therapeutic options were available to extend survival or for which the participant was not a candidate for standard-of-care therapy.
3. Eastern Cooperative Oncology Group performance status ≤ 1.
4. Life expectancy ≥ 3 months.
5. ≥ 1 injectable, measurable (≥ 10 mm in diameter, or ≥ 15 mm for nodal lesions), eligible lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Eisenhauer et al 2009), immune-related RECIST (iRECIST) (Seymour et al 2017), and/or Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) (Cheson et al 2016) and as assessed by the Investigator. Eligible lesions must not have been located in the thoracic cavity, spleen, pancreas, gastrointestinal tract (liver injection allowed), or cranium and must have been amenable to percutaneous injection and away from major blood vessels or neurological structures.
6. Able to provide biopsies for biomarker analysis from injected and (if available) noninjected lesions at baseline and other time points during the study.
7. Oxygen saturation > 90% without the use of supplemental oxygen.
8. Adequate cardiac function, defined as follows:

   1. Left ventricular ejection fraction (LVEF) > 50% by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO) performed within 6 months prior to the first dose of study treatment provided the participant had not received any potential cardiotoxic agents in the intervening period. Symptoms relating to left ventricular dysfunction, cardiac arrhythmia, or cardiac ischemia must all have been Grade < 1 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
   2. QTc interval corrected for heart rate using Fridericia's formula (QTcF) < 480 msec at screening.
9. Laboratory values within the following ranges:

   * Absolute neutrophil count ≥ 1500/µL
   * Lymphocyte count ≥ 500/µL
   * Platelets ≥ 100,000/µL without transfusion
   * Hemoglobin ≥ 9.0 g/dL (participants may have been transfused to meet this criterion)
   * Estimated glomerular filtration rate (eGFR) > 50 mL/min/1.73 m^2 per the Cockcroft-Gault formula
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN or ≤ 3 × ULN for participants with Gilbert's syndrome
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 × ULN (AST and ALT ≤ 5 × ULN for participants with liver metastases and alkaline phosphatase ≤ 5 × ULN for participants with liver or bone metastases)
   * International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant was receiving anticoagulant therapy as long as PT or aPTT was within therapeutic range of intended use of anticoagulants
10. Agreed to use an acceptable method of contraception after informed consent, throughout the study, and for 5 months after the last dose of SYNB1891 or atezolizumab.

    Additional inclusion criteria that applied only to Arm 2 study participants were as follows:
11. Thyroid-stimulating hormone (TSH) within the normal reference range or the participant was receiving stable thyroid replacement therapy.
12. Participants must have received treatment with an anti-programmed cell death protein-1 (PD-1)/programmed death-ligand 1 (PD-L1) monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors (CPIs) or other therapies, if indicated (if CPI therapy was not indicated as a part of standard-of-care therapy, participants may have been CPI naïve).

Exclusion Criteria

1. Chemotherapy, radiation, or biological cancer therapy within 14 days prior to the first dose of study treatment, or failure of any adverse events (AEs) to recover to Baseline or NCI CTCAE version 5.0 Grade 1, except for any grade of alopecia caused by cancer therapeutics administered > 28 days earlier.
2. Systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 28 days or 5 drug elimination half-lives (whichever was longer) prior to initiation of study treatment. CPIs were not considered systemic immunostimulatory agents for this criterion and were subject to the washout period listed in exclusion criterion #1.
3. Allogeneic hematopoietic stem cell transplantation that required current use of immunosuppressors.
4. Receipt of a live vaccine within 90 days prior to the first dose of study treatment or anticipation of a need for such a vaccine during treatment.
5. Receipt of antibiotics within 7 days prior to the first dose of study treatment.
6. Participation in a study of an investigational agent and receipt of study therapy or use of an investigational device within 28 days prior to the first dose of study treatment.
7. Diagnosed immunodeficiency or current use of chronic systemic steroid therapy in excess of replacement doses (prednisone ≤ 10 mg/day or equivalent was acceptable) or any other form of immunosuppressive medication within 7 days prior to the first dose of study treatment.
8. For injection and biopsy of visceral (deep) lesions: participants must not have been on long-acting antiplatelet agents such as aspirin or clopidogrel or on therapeutic doses of anticoagulants, with the exception of participants receiving a preventative dose of low molecular weight heparin. In participants receiving preventative low molecular weight heparin, treatment must have been stopped 24 hours before the intratumoral injection and resumed again 24 hours after the injection (Marabelle et al 2018).
9. Previous or concurrent malignancy, with the exception of:

   1. Adequately treated basal or squamous cell carcinoma, in situ carcinoma of the cervix, or ductal carcinoma in situ of the breast;
   2. Localized prostate cancer definitively treated with surgery or radiation or stable on hormone therapy;
   3. Other cancer from which the participant had been disease free for at least 2 years.
10. Clinically active central nervous system metastases and/or carcinomatous meningitis (treated brain metastases were permitted if radiologically stable for ≥ 28 days prior to the first dose of study treatment).
11. Allergy to antibiotics that precluded treatment for infection with Escherichia coli Nissle 1917.
12. Hepatitis B or C infection(s) unless screening tests indicated a negative viral load, and/or human immunodeficiency virus infection unless screening tests indicated a negative or below the limit of quantitation viral load.
13. Known active tuberculosis.
14. Grade 3 or higher infection according to NCI CTCAE within 28 days prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
15. Failure to fully recover from the effects of major surgery. Surgeries that required general anesthesia must have been completed > 14 days before the first dose of study drug. Surgery requiring regional/epidural anesthesia must have been completed > 72 hours before the first dose of study treatment and participants should have recovered.
16. Heart failure of New York Heart Association Class 3 or greater, restrictive cardiomyopathy, or unstable angina or recent myocardial infarction within 3 months prior to the first dose of study treatment.
17. Any other medical condition that might have confounded the results of the study, interfered with the participant's participation, or was not in the best interest of the participant, in the opinion of the treating Investigator.
18. Pregnant or breastfeeding or anticipated conception or fathering of children within the projected duration of the study and for 5 months after the last dose of SYNB1891 or atezolizumab.

    Additional exclusion criteria that applied only to Arm 2 study participants were as follows:
19. History of immune-mediated AEs on prior PD-1/PD-L1 therapies requiring discontinuation or immunosuppressor therapy, excluding endocrinopathies.
20. Active or history of underlying autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    1. Participants with a history of autoimmune-related hypothyroidism who were on thyroid replacement hormone were eligible for the study.
    2. Participants with controlled Type 1 diabetes mellitus who were on an insulin regimen were eligible for the study.
    3. Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis are excluded) were eligible for the study provided all of following conditions were met:

       * Rash covered < 10% of body surface area;
       * Disease was well controlled at baseline and required only low potency topical corticosteroids;
       * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
21. History of a Grade ≥ 3 allergic anaphylactic reaction following treatment with a PD-1 mAb or to chimeric, human, or humanized antibodies or fusion proteins.
22. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis requiring treatment, or idiopathic pneumonitis, or evidence of active pneumonitis.
23. Known hypersensitivity to Chinese hamster ovary cell products or any component of the atezolizumab formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aoife Brennan, MB, BCh, BAO, MMSc, Study Director — Synlogic
Locations (6):
- United States (6):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Hackensack University John Theurer Cancer Center, Hackensack, New Jersey
  - Ohio State University College of Medicine, Columbus, Ohio
  - University of Pittsburgh Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Cheson BD, Ansell S, Schwartz L, Gordon LI, Advani R, Jacene HA, Hoos A, Barrington SF, Armand P. Refinement of the Lugano Classification lymphoma response criteria in the era of immunomodulatory therapy. Blood. 2016 Nov 24;128(21):2489-2496. doi: 10.1182/blood-2016-05-718528. Epub 2016 Aug 29. PMID 27574190
- [Background] Ji Y, Wang SJ. Modified toxicity probability interval design: a safer and more reliable method than the 3 + 3 design for practical phase I trials. J Clin Oncol. 2013 May 10;31(14):1785-91. doi: 10.1200/JCO.2012.45.7903. Epub 2013 Apr 8. PMID 23569307
- [Background] Marabelle A, Andtbacka R, Harrington K, Melero I, Leidner R, de Baere T, Robert C, Ascierto PA, Baurain JF, Imperiale M, Rahimian S, Tersago D, Klumper E, Hendriks M, Kumar R, Stern M, Ohrling K, Massacesi C, Tchakov I, Tse A, Douillard JY, Tabernero J, Haanen J, Brody J. Starting the fight in the tumor: expert recommendations for the development of human intratumoral immunotherapy (HIT-IT). Ann Oncol. 2018 Nov 1;29(11):2163-2174. doi: 10.1093/annonc/mdy423. PMID 30295695
- [Derived] Luke JJ, Piha-Paul SA, Medina T, Verschraegen CF, Varterasian M, Brennan AM, Riese RJ, Sokolovska A, Strauss J, Hava DL, Janku F. Phase I Study of SYNB1891, an Engineered E. coli Nissle Strain Expressing STING Agonist, with and without Atezolizumab in Advanced Malignancies. Clin Cancer Res. 2023 Jul 5;29(13):2435-2444. doi: 10.1158/1078-0432.CCR-23-0118. PMID 37227176

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells): SYNB1891 was administered as an intratumoral (IT) injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles.
- Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells); Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells); Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells); Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells); Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells): SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles.
- Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab: SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles in combination with standard dose atezolizumab (1200 mg intravenously [IV] every 3 weeks [Q3W]) on Day 1 of each cycle.
- Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab: SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles in combination with standard dose atezolizumab (1200 mg IV Q3W) on Day 1 of each cycle.
Period: Overall Study
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab
Started | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4
Completed (Defined as completing treatment with study drug(s) for four 21-day cycles) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 5 | 2 | 6 | 4 | 4
Not completed — Disease progression | 1 | 1 | 3 | 3 | 2 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled, allocated to treatment, and received at least 1 dose of investigational product.
Groups:
- Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells); Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells); Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells); Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells); Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells); Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells): SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles.
- Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab; Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab: SYNB1891 was administered as an IT injection on Days 1, 8, and 15 of Cycle 1 and Day 1 of subsequent cycles in combination with standard dose atezolizumab (1200 mg IV Q3W) on Day 1 of each cycle.
- Total: Total of all reporting groups
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab | Total
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 21
  >=65 years | 1 | 0 | 1 | 2 | 0 | 5 | 1 | 1 | 11
Age, Continuous [Median (Full Range); unit: years] | 62.0 [25 to 68] | 58.0 [51 to 61] | 53.5 [46 to 70] | 57.0 [43 to 79] | 63.0 [60 to 63] | 74.5 [53 to 82] | 59.5 [37 to 74] | 60.5 [54 to 77] | 61.5 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 4 | 1 | 4 | 2 | 1 | 20
  Male | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 4 | 5 | 3 | 6 | 3 | 4 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  White | 2 | 3 | 3 | 5 | 3 | 5 | 4 | 4 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4 | 32
Disease type [Count of Participants; unit: Participants]
  Melanoma | 1 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 8
  Sarcoma | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 5
  Esophageal cancer | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4
  Squamous cell carcinoma (oropharynx) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Ampullary bile duct adenocarcinoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Basal cell carcinoma | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cecum adenocarcinoma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Colorectal cancer | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Endometrial cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Jejunum adenocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Merkel cell carcinoma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Non-small cell lung cancer | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Rectosigmoid adenocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Small cell lung cancer | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Squamous cell carcinoma (skin) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Squamous cell carcinoma (vulva) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Testicular cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity
Description: The following adverse events (AEs) were DLTs if they occurred in Cycle 1 and were assessed by the Investigator as related to treatment:
  1. Grade (Gr) 4 nonhematologic toxicity (not laboratory)
  2. Gr 4 hematologic toxicity ≥ 7 days, any Gr 4 thrombocytopenia, or Gr 3 thrombocytopenia with significant bleeding
  3. Gr ≥ 3 nonhematologic toxicity (exceptions: Gr 3 fatigue ≤ 3 days; Gr 3 diarrhea, nausea, or vomiting without treatment; Gr 3 rash without treatment)
  4. Gr 3/4 nonhematologic laboratory value for > 1 week or resulting in significant medical intervention, hospitalization, or drug-induced liver injury (exceptions: clinically nonsignificant, treatable, or reversible laboratory abnormalities)
  5. Gr 3/4 febrile neutropenia
  6. Sepsis, severe abscesses and/or ulcerations requiring surgical management
  7. Toxicity delaying Cycle 2 initiation >2 weeks
  8. Toxicity causing treatment discontinuation
  9. Gr 3 toxicity causing omission of > 33% of study doses
  10. Gr 5 toxicity
Time Frame: 21 days (1 cycle)
Population: All participants who were enrolled, allocated to treatment, and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) vs Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) vs Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) vs Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) vs Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) vs Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) vs Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab vs Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab; Because only 1 participant experienced a DLT (Grade 3 cytokine release syndrome in Arm 1 Cohort 6), no MTD could be reached; Test type: Other; Because only 1 participant experienced a DLT (Grade 3 cytokine release syndrome in Arm 1 Cohort 6), no MTD could be reached

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, as follows: Grade 1 (mild/asymptomatic; no intervention); Grade 2 (moderate; minimal intervention); Grade 3 (severe/medically significant; hospitalization indicated; disabling); Grade 4 (life-threatening; urgent intervention required); or Grade 5 (fatal). Adverse events (AEs) were reported from clinical laboratory tests, vital sign and weight measurements, physical examinations, and any other medically indicated assessments, including participant interviews, from the time informed consent was signed through the end of the safety follow-up period. AEs were considered to be treatment-emergent adverse events (TEAEs) if they occurred or worsened in severity after the first dose of study treatment. TEAEs were considered treatment-related if the relationship to study drug was possibly, probably, or definitely related.
Time Frame: Up to 13 months
Population: All participants who were enrolled, allocated to treatment, and received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab
Number analyzed (Participants) | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4
Participants
  Any TEAE | 3 | 3 | 4 | 5 | 3 | 6 | 4 | 4
  Maximum TEAE severity Grade 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
  Maximum TEAE severity Grade 2 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 1
  Maximum TEAE severity Grade 3 | 1 | 0 | 1 | 3 | 1 | 3 | 0 | 1
  Maximum TEAE severity Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum TEAE severity Grade 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  TEAE related to SYNB1891 | 3 | 1 | 2 | 3 | 3 | 6 | 2 | 2
  TEAE related to atezolizumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  TEAE leading to treatment withdrawal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Best Tumor Response as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: Appropriate imaging of the SYNB1891-injected tumor(s) and up to 5 target (noninjected) lesions was performed at baseline and every 2 cycles during the treatment period. Tumor response was assessed by the local investigator using RECIST 1.1 (Eisenhauer et al 2009). Per RECIST 1.1, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 13 months
Population: All participants who received study drug and had an on-treatment response assessment (including "Not Evaluable") or who discontinued study before any response assessment was performed due to disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 3 | 3 | 4 | 3
Participants
  SD | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2
  PD | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time a participant signed informed consent through the safety follow-up period were documented, regardless of the causal relationship to study drug. AEs that occurred or worsened in severity after the first dose of study treatment were considered treatment emergent (i.e., TEAEs). The longest duration of study participation for any participant was 13 months.
Description: AE documentation included duration (onset and resolution dates), severity using the NCI CTCAE (version 5.0), assessment of causality, seriousness, and whether specific action or therapy was required. In summaries, preferred terms are counted only once per participant at the maximum reported grade.
Arm/Group | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 0/4 | 1/5 | 0/3 | 0/6 | 0/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/4 | 3/5 | 0/3 | 3/6 | 0/4 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 5/5 | 3/3 | 6/6 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) (N=3) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) (N=3) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) (N=4) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) (N=5) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) (N=3) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) (N=6) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab (N=4) | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab (N=4)
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovial sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Cohort 1: SYNB1891 Monotherapy (1 × 10^6 Live Cells) (N=3) | Arm 1 Cohort 2: SYNB1891 Monotherapy (3 × 10^6 Live Cells) (N=3) | Arm 1 Cohort 3: SYNB1891 Monotherapy (1 × 10^7 Live Cells) (N=4) | Arm 1 Cohort 4: SYNB1891 Monotherapy (3 × 10^7 Live Cells) (N=5) | Arm 1 Cohort 5: SYNB1891 Monotherapy (1 × 10^8 Live Cells) (N=3) | Arm 1 Cohort 6: SYNB1891 Monotherapy (3 × 10^8 Live Cells) (N=6) | Arm 2 Cohort 1: SYNB1891 (1 × 10^7 Live Cells) + Atezolizumab (N=4) | Arm 2 Cohort 2: SYNB1891 (3 × 10^7 Live Cells) + Atezolizumab (N=4)
Chills (General disorders) | 1 | 1 | 0 | 1 | 2 | 4 | 2 | 2
Pyrexia (General disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Corona Virus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Uric Acid Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discharge (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the Sponsor prior to enrollment completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT04167137/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04167137/SAP_001.pdf